CLINICAL TRIAL: NCT05125497
Title: Natural Cycle, Minimal Stimulation and Conventional IVF: a Registry-based Comparison of the IVF Treatments, Their Efficacy and Pregnancy Outcomes
Brief Title: Natural Cycle, Minimal Stimulation and Conventional IVF: a Registry-based Study
Acronym: IVF-Regsitry
Status: Completed | Type: Observational
Sponsor: Universitätsklinik fur Frauenheilkunde, Inselspital Bern (Other)
Responsible Party: Principal Investigator, Magaton Isotta, Dr. med. Isotta Martha Magaton, Universitätsklinik fur Frauenheilkunde, Inselspital Bern
Other Study IDs: 2021-01689 (BASEC-ID); LB1562_NC-IVF (Other: RedCap ID); Study Number 4949 (Other: Department Lehre und Forschung Inselspital Bern)
Record Dates: First submitted 2021-11-03; First posted 2021-11-18 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: IVF
MeSH Terms: interventions — Fertilization in Vitro

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- In Vitro Fertilisation (IVF)-Patients: Patients aim to do In-Vitro-Fertilisation (IVF)
  Interventions: Procedure: In Vitro Fertilisation (IVF)

INTERVENTIONS:
Procedure: In Vitro Fertilisation (IVF) — Natural Cycle In Vitro Fertilisation (IVF): without hormonal stimulation Conventional In Vitro Fertilisation (IVF): conventional hormonal stimulation Minimal Stimulation In Vitro Fertilisation (IVF): low dose of hormonal stimulation will be applied

SUMMARY:
International prospective registry-based study of different types of In Vitro Fertilisation (IVF) and their outcome.

DETAILED DESCRIPTION:
One year of prospective collection of descriptive In-Vitro-Fertilisation data. The data will be collected in 13 In-Vitro-Fertilisation-centres

ELIGIBILITY:
Inclusion criteria: In Vitro Fertilisation and signed informed consent

Exclusion criteria:

* Medical freezing
* Social freezing
* thawed cycles

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — women
Study Population: Patients aiming to do In Vitro Fertilisation with fresh embryo transfer
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Implantation rate | 1 year
  pregnancy rate per transferred embryo

SECONDARY OUTCOMES:
Number of oocytes | 1 Year
  Number of retrieved oocytes per protocol
Clinical pregnancy rate | 1 year
  Pregnancy rate per transfer
Pregnancy outcome | 1 year
  Pregnancy complications including preeclampsia
In Vitro Fertilisation complications rates | 1 year
  miscarriage

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsfrauenklinik Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Magaton IM, Siercks I, Nordin M, Popovici RM, Boogen EM, Eisenhardt S, Reeka N, Lanowski JS, Roumet M, von Wolff M. Oocyte and zygote development potential in minimal stimulation, natural cycle and conventionally stimulated IVF: an international multi-centre retrospective cohort study. J Assist Reprod Genet. 2025 Jul;42(7):2331-2340. doi: 10.1007/s10815-025-03508-3. Epub 2025 May 28. PMID 40434705